CLINICAL TRIAL: NCT02825706
Title: Effectiveness of an Educational Physiotherapy and Home Exercises Program in Adult Patients With Hemophilia: A Randomized Clinical Trial
Brief Title: Educational Physiotherapy in Haemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Fundación Victoria Eugenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EducationalPhys
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Haemophilia
Keywords: Hemophilia; Educational Physiotherapy; Pain; Quality of life; Illness Behaviour; Elbow
MeSH Terms: conditions — Hemophilia A; Pain; Illness Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): The patients in experimental group received 60-minute educational sessions every two weeks about the pathophysiology of hemophilia, clinical manifestations, postural advice and prevention advice to avoid recurrent bleeding. Likewise, doubts on the clinical progress of hemophilic arthropathy, functional limitations and management of joint pain were resolved. In parallel with the educational sessions, patients followed a 15-week home exercise program performed once a day, 6 days a week. The program included muscle stretching exercises; isometric exercises; proprioceptive exercises on one leg with visual support; and a 20-minute walk. Low-intensity exercises with 20-25 repetitions were included.
  Interventions: Other: Educational physiotherapy group
- Control group (No Intervention): The patients in the control group did not receive any educational sessions and did no exercise at all at home.

INTERVENTIONS:
Other: Educational physiotherapy group — 20 patients with hemophilia were randomly allocated to an educational intervention or to a control group. The educational intervention was performed every two weeks during 15-week and home exercises were performed once a day, 6 days a week, in the same time
  Arms: Experimental group

SUMMARY:
Although arthropathy is a serious problem in patients with hemophilia due to the associated morbidity and incapacity, to the best of the investigators knowledge, no studies have looked at the effect of educational physiotherapy for its clinical improvement.

This contribution presents the results of educational physiotherapy program applied for 15 weeks with home exercises - in patients with hemophilic arthropathy. After treatment, experimental group showed improved a significant reduction of pain, and best quality of life al illness behaviour. During treatment no patient showed elbow haemarthrosis, which underlines the safety of this physiotherapy program.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A or B
* Patients over 18 years
* Patients with hemophilic arthropathy with at least 1 involved joint (elbow, knee or ankle)
* having signed the informed consent document.

Exclusion Criteria:

* Patients diagnosed with other congenital bleeding disorders (i.e. von Willebrand disease)
* Patients who developed antibodies to FVIII or FIX (inhibitors)
* Those not able to ambulate as a result of hemophilic arthropathy or any other disability

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline physical condition of joints after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  The physical condition of joints was assessed using the Gilbert scale that measures swelling, muscle atrophy, joint crepitus, range of motion, axial deformity and instability. Scores range from 0 to 12 (0 represents no joint injury and 12 represents maximum joint deterioration).
Change from baseline joint pain after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  Joint pain was assessed using the Visual Analog Scale (VAS), with scores ranging from 0 (no pain at all) to 10 (the worst pain imaginable by the patient).
Change from baseline perception of the quality of life after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  The Haemophilia A-36 questionnaire was used to assess the perception of the quality of life. This questionnaire consists of 36 items that assess 9 domains (physical health, daily activities, joint damage and pain, treatment satisfaction, treatment difficulties, emotional functioning, mental health and social relationships).
Change from baseline illness behavior after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  To assess illness behavior, patients completed the Illness Behavior Questionnaire (IBQ). This scale consists of 62 items and 8 domains (hypochondriasis, disease conviction, psychological vs. somatic perception of illness, affective inhibition, affective disturbance, denial and irritability).
Change from baseline frequency of bleedings after treatment and at 6 months | Screening visit, within the first seven days after treatment and after six months follow-up visit
  The frequency of bleeding is measured with a record which complete the patients, where they indicate the incidence of hematomas and hemarthrosis during the treatment and follow-up.

SECONDARY OUTCOMES:
Radiological joint deterioration | Screening visit
  All patients had an assessment of radiological joint deterioration using the Pettersson scale. This scale, with scores ranging from 0 (a normal joint) to 13 (maximum joint deterioration), is the most widely used to assess joint degeneration produced by hemophilic arthropathy. The evaluation of radiological joint damage was done at the beginning of the study.
Age | Screening visit
  Age of patients included in the study
Weight | Screening visit
  Weight of the patients
Height | Screening visit
  Height of patients

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Real Fundación Victoria Eugenia

IPD SHARING:
Plan to Share IPD: No